CLINICAL TRIAL: NCT05105399
Title: Evaluation of Serratus Plane Block on the Respiratory Pattern in Patients With Multiple Rib Fractures: a Perspective Randomized Controlled Study
Brief Title: Evaluation of Serratus Plane Block on the Respiratory Pattern in Patients With Multiple Rib Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP Versione 2 del 05/06/2020
Record Dates: First submitted 2021-10-20; First posted 2021-11-03 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Rib Fractures; Spirometry
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morphine (No Intervention)
- Continuous (Active Comparator)
  Interventions: Procedure: Serratus plane block (continuous or single-shot)
- Single (Active Comparator)
  Interventions: Procedure: Serratus plane block (continuous or single-shot)

INTERVENTIONS:
Procedure: Serratus plane block (continuous or single-shot) — Patients assigned to the interventional arms will receive either continuous serratus plane block or single-shot serratus plane block
  Arms: Continuous; Single

SUMMARY:
In patients admitted following a trauma, the incidence of multiple rib fractures is reported to be 9,7%, and this can be even higher in high energy trauma like motor vehicle accidents (1). Pain deriving from rib fractures cause the patient to breath shallow in order to limit discomfort and this bring about negative consequences: shallow breathing and inability to clear secretions may cause pulmonary atelectasis eventually evolving to pneumonia. Given the aforementioned concerns, it is easy to understand why, in a context like this, control of chest pain become crucial. The best way to achieve adequate pain control have not yet been established: the aim of this study is to investigate on this clinical dilemma. In this study, 72 people with at least two monolateral rib fractures are going to be randomized into three groups: 1) standard treatment alone (intravenous analgesia: acetaminophen + morphine PCA); 2) continuous serratus plane block + standard treatment; 3) single-shot serratus plane block + standard treatment. The variables that are going to be recorded are the following: pain through the NRS scale, FEV1 and FVC through spirometry and finally an arterious gas analysis. Recording are going to be repeated at 72h after admission. The primary endpoint is to evaluate if the continuous serratus plane block is able to improve the FEV1/FVC compared to single shot or standard treatment alone. Secondary endpoints will be: the effect of continuous block on 1) resting and incident pain; 2) opioid consumption; 3) blood gas analysis parameters; 4) pulmonary complications at 1 month; 5) length of stay

ELIGIBILITY:
Inclusion Criteria:

1. Chest trauma with at least 2 monolateral rib fractures (monofocal or multifocal) with no flail chest
2. Age>18 years
3. Hospital admission
4. Ability to provide written informed consensus
5. Awake patient, spontaneous ventilation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
FEV1 (% of the predicted value) | 72 hours
  Any statistically significant difference between the two treatment groups and the control group will be measured. FEV1 is expected to be respectively 80±15% of the predicted value in the treatment groups and 64±15% of the predicted value in the control group

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided